CLINICAL TRIAL: NCT02681185
Title: Efficacy of a Virtual Care Clinic in the Management of Diabetes Mellitus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment not satisfied
Sponsor: Endocrine Research Society (Other)
Responsible Party: Principal Investigator, ERS Gap Student, Clinical Professor, Endocrine Research Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Virtual Care
Record Dates: First submitted 2016-01-19; First posted 2016-02-12 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Telemedicine; Standard of Care

STUDY DESIGN:
Intervention Model Description: Experimental vs. Standard of Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): The recruited participants will be provided access to Virtual Care suite via internet and telephone communication.
  Interventions: Other: Virtual Care
- Standard of Care (Active Comparator): The recruited participants will receive the standard of diabetes care as offered by the services in their community.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Virtual Care — Virtual Care consists of the following services and resources:
  1. Have a virtual consult through online methods or telephone with one of the study endocrinologists
  2. Be encouraged to report blood sugar readings every 2 weeks to their endocrinologist for regular follow-up and feedback via online methods
  3. Be given access to a website with modules that attempt to replicate the information learned in a diabetes teaching clinic
  4. Be given access to a certified diabetes educator through online methods or telephone. This will cover any other information that cannot be personalized on the teaching website, such as specific diet advice and social support.
  Arms: Interventional Group
Other: Standard of Care — Standard of care offered in the patient's community. May involve in-person education at a diabetes centre and consultation with a healthcare professional.
  Arms: Standard of Care

SUMMARY:
The study's goal is to promote accessible and cost-effective diabetes care through electronic means. Underserved populations including rural areas do not have diabetes specialists. Previous study data has shown the effectiveness of Internet communication in lowering a patient's Hemoglobin A1C, a measure of blood sugars, closer to the target number. The investigators thus wish to test the effectiveness of diabetes care provided by virtual means, including virtual consultations, online monitoring of blood sugars, diabetes education via web-based videos, and support/advice provided through phone or email by an Endocrinologist. The goal is to test if virtual care is a viable means to extend care for diabetes to underserved populations.

DETAILED DESCRIPTION:
1. Purpose To determine if a virtual-care based system can effectively provide care for patients with diabetes.
2. Hypothesis Alternative: Virtual-care is associated with achieving glycemic control in patients with diabetes.

   Null: Virtual-care is not associated with achieving glycemic control in patients with diabetes.
3. Justification The potential study participants would normally receive care from a primary care physician and have no access to a diabetes specialist. In the study, they would have access to an Endocrinologist through online communication and by telephone.
4. Objectives The primary end-point is to determine if patients using virtual care have reduced HbA1c values at followup. The data may be used to write a white paper guiding diabetes treatment guidelines within the province of British Columbia, Canada. The goal is for diabetes specialists to be able to provide care to underserved areas without requiring to be physically at the location.
5. Research Method Participants satisfying the inclusion criteria will be recruited and followed for six months. Their family physician or Diabetes Center will provide a referral to one of the investigators, who are diabetes specialists, for a virtual consult via telephone. Relevant medical records will be transferred for this consult.

   After the consult, participants will be asked to submit self-monitored blood glucose levels via email to the diabetes specialists for follow-up every two weeks. These follow-up reports may lead to the diabetes specialists making adjustments to therapy.

   Concurrently, the participants during the followup period will be provided access to a free website containing modules on diabetes education similar to a diabetes clinic education program. They will be allowed to view them at their own discretion..

   Every 3 months participants will be asked to have regular blood work done to assess management, including A1C levels. This is part of routine care, but the data will be used for analysis.
6. Statistical Analysis Outcomes will be tested for significant differences via t tests, as well as the other clinical measures, while the summarized survey responses will be tallied and tested for correlation with changes in clinical measures.

The planned sample size of 100 was estimated from previous studies' mean changes in A1C and standard deviations involving similar methods. For calculating the sample size, a statistical power of 0.80 and alpha of 0.05 were used.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Access and the ability to use the internet on a computer or mobile device
* Access to a family physician and lab for blood tests

Exclusion Criteria:

* Patients that are pregnant or attempting to conceive
* Liver disease (AST or ALT levels >2.5 times the reference level)
* Renal insufficient with a serum creatine level >200 umol/L
* Patients who see an endocrinologist or diabetes specialist within their community

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 month intervals for 6 months
  Routine blood work measuring average blood sugar levels, at total of two tests will be preformed at three month intervals over the 6 month study period. Baseline A1C at recruitment will also be included in analysis.

SECONDARY OUTCOMES:
Survey of Healthcare Utilization | Start and End of study (six months)
  At the start and end of study (six months), participants will complete a self-reported survey of their utilization of healthcare services, including hospitalizations, physician visits, intervention website visits, perceived medication changes.
Survey of Quality of Life | Start and End of study (six months)
  At the start and end of study (six months), participants will complete the Audit for Diabetes Dependent Quality of Life survey.

CONTACTS AND LOCATIONS:
Overall Officials: Adam White, MD, Principal Investigator — Clinical Associate Professor, UBC; Monika Pawlowska, MD, Principal Investigator — Clinical Assistant Professor, UBC
Locations (1):
- Endocrine Research Society, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Data collected during the study will be stored on study site in an encrypted format, all data pertaining to individual patients will be available only to the study investigators.

REFERENCES:
- [Background] Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, Raskin P, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;353(25):2643-53. doi: 10.1056/NEJMoa052187. PMID 16371630
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Hirsch IB, Bode BW, Childs BP, Close KL, Fisher WA, Gavin JR, Ginsberg BH, Raine CH, Verderese CA. Self-Monitoring of Blood Glucose (SMBG) in insulin- and non-insulin-using adults with diabetes: consensus recommendations for improving SMBG accuracy, utilization, and research. Diabetes Technol Ther. 2008 Dec;10(6):419-39. doi: 10.1089/dia.2008.0104. PMID 18937550
- [Background] Austin MM, Haas L, Johnson T, Parkin CG, Parkin CL, Spollett G, Volpone MT. Self-monitoring of blood glucose: benefits and utilization. Diabetes Educ. 2006 Nov-Dec;32(6):835-6, 844-7. doi: 10.1177/0145721706295873. No abstract available. PMID 17102152
- [Background] Tildesley HD, Mazanderani AB, Ross SA. Effect of Internet therapeutic intervention on A1C levels in patients with type 2 diabetes treated with insulin. Diabetes Care. 2010 Aug;33(8):1738-40. doi: 10.2337/dc09-2256. PMID 20668152
- [Background] Tildesley HD, Wright AM, Chan JH, Mazanderani AB, Ross SA, Tildesley HG, Lee AM, Tang TS, White AS. A comparison of internet monitoring with continuous glucose monitoring in insulin-requiring type 2 diabetes mellitus. Can J Diabetes. 2013 Oct;37(5):305-8. doi: 10.1016/j.jcjd.2013.05.006. PMID 24500556
- [Background] Tildesley HD, Conway ME, Ross SA, Lee AM, Chan JH, Mazanderani AB, Tildesley HG, White AS. Review of the effect of internet therapeutic intervention in patients with type 1 and type 2 diabetes. Diabetes Care. 2014 Feb;37(2):e31-2. doi: 10.2337/dc13-1940. No abstract available. PMID 24459161
- [Background] Tildesley HD, Po MD, Ross SA. Internet blood glucose monitoring systems provide lasting glycemic benefit in type 1 and 2 diabetes: a systematic review. Med Clin North Am. 2015 Jan;99(1):17-33. doi: 10.1016/j.mcna.2014.08.019. Epub 2014 Oct 18. PMID 25456641